CLINICAL TRIAL: NCT02927184
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Assess The Efficacy, Safety, and Tolerability of VK2809 Administered for 12 Weeks Followed by a 4-Week Off-Drug Phase in Patients With Primary Hypercholesterolemia and Non-Alcoholic Fatty Liver Disease
Brief Title: Safety and Tolerability of VK2809 in Patients With Primary Hypercholesterolemia and Non-Alcoholic Fatty Liver Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Viking Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VK2809-201
Record Dates: First submitted 2016-10-05; First posted 2016-10-06 (Estimated); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Hyperlipidemia; NAFLD
MeSH Terms: conditions — Hyperlipidemias; Non-alcoholic Fatty Liver Disease | interventions — 2-((3,5-dimethyl-4-(4'-hydroxy-3'-isopropylbenzyl)phenoxy)methyl)-4-(3-chlorophenyl)-2-oxido(1,3,2)dioxaphosphonane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Placebo capsule
  Interventions: Drug: Placebo
- VK2809 (5mg) (Experimental): 5mg VK2809 capsule
  Interventions: Drug: VK2809
- VK2809 (10mg) (Experimental): 10mg VK2809 capsule
  Interventions: Drug: VK2809
- VK2809 (10mg QOD) (Experimental): 10mg VK2809 capsule
  Interventions: Drug: VK2809

INTERVENTIONS:
Drug: VK2809
  Arms: VK2809 (10mg QOD); VK2809 (10mg); VK2809 (5mg)
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will investigate the efficacy, safety, and tolerability of VK2809 in lowering LDL-C and liver fat content in patients with primary hypercholesterolemia and fatty liver disease. The primary efficacy endpoint is percent change from baseline LDL-C at the end of the treatment period (Week 12). Secondary endpoints include effects on liver fat content and other liver and lipid markers, as well as effects on safety and tolerability, and pharmacokinetic (PK) measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Minimum of 10% liver fat as assessed by MRI - Proton Density Fat Fraction
2. Fasting serum LDL-C >130 mg/dL at screening, >110 mg/dL on lipid lowering medications
3. Any one of the following:

   1. Triglycerides ≥150 mg/dL or receiving prescription medication for elevated triglycerides.
   2. Systolic blood pressure >130 mmHg or diastolic blood pressure ≥85 mmHg or receiving prescription medication for hypertension.
   3. Waist circumference >40 inches (men) or >35 inches (women)
4. Body mass index (BMI) 18.50 - 40.00 kg/m2 inclusive at screening
5. Provide a personally-signed and dated informed consent document

Exclusion Criteria:

1. Females of childbearing potential and males unwilling to use barrier birth control method (condom) throughout the study
2. Resting 12-lead ECG showing QTc >450 msec, any tachyarrhythmia or morphology change, or any other clinically significant abnormality
3. Cardiovascular event requiring hospitalization in the past year
4. History or presence of thyroid disorder
5. History of malignancy in past 5 years
6. LDL-C ≥190 mg/dL or familial hypercholesterolemia
7. Significant hepatic or renal function test abnormalities

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2016-09-28 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
Change in LDL-C in patients receiving VK2809 compared to placebo | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Mancini, Study Director — Viking Therapeutics, Inc.
Locations (17):
- United States (17):
  - Radiant Research, Inc., Chandler, Arizona
  - SC Clinical Research, Garden Grove, California
  - ACTCA, Los Angeles, California
  - Catalina Research Institute, Montclair, California
  - North America Research, Inc, Pomona, California
  - Orange County Research Center, Tustin, California
  - Research Institute of South Florida, Miami, Florida
  - Avant Research Associates, LLC, Crowley, Louisiana
  - HCI- MetroMedic Walk-in, New Bedford, Massachusetts
  - Flint Clinical Research, PLLC, Flint, Michigan
  - Mid Hudson Medical, Hopewell Junction, New York
  - CHEAR Center, LLC, The Bronx, New York
  - Wake Research Associcates, LLC., Raleigh, North Carolina
  - Avant Research, Beaumont, Texas
  - Clinical Trials of Texas, INC, San Antonio, Texas
  - Radiant Research, Inc., San Antonio, Texas
  - Wasatch Clinical Research, LLC, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No